CLINICAL TRIAL: NCT00253864
Title: Functional Outcome Following Shoulder Surgery: A Prospective Database
Brief Title: Functional Outcomes Following Shoulder Surgery: A Prospective Database
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2003658-01H
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Rotator Cuff Tear
Keywords: shoulder surgery; prospective database; long term outcome
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arthroscopic rotator cuff repair: Participants who underwent an arthroscopic rotator cuff repair between 2007-2009.
  Interventions: Procedure: Single row; Procedure: Double row

INTERVENTIONS:
Procedure: Single row — Fixation type in arthroscopic rotator cuff repair.
Procedure: Double row — Fixation type in arthroscopic rotator cuff repair.

SUMMARY:
The purpose of this prospective database is to investigate the long-term functional status of patients who have undergone various types of rotator cuff repair surgery. Patients are asked to respond to questionnaires prior to surgery and at various post-operative visits in an attempt to quantify their functional outcomes. Responses are then linked to other data such as symptoms, prior treatments, previous surgery, complications, radiographic results, etc. These data may then be used as a basis for devising guidelines for future patients and surgeons. This particular project is interested in investigating long term results of arthroscopic rotator cuff repair techniques.

DETAILED DESCRIPTION:
The purpose of the prospective database is to initiate data collection for a group of patients undergoing surgery of the shoulder. Long-term data collection will include information on the functional status of the patients' shoulder as well as quality of life information and radiographic results.

For the purposes of this study, we are interested in the long-term outcomes of participants who underwent a double row versus single row fixation in arthroscopic rotator cuff repair procedures.

ELIGIBILITY:
Inclusion Criteria:

* arthroscopic rotator cuff repairs that occurred between 2007-2009
* enrolled in previous study comparing single vs double-row fixation

Exclusion Criteria:

* withdrew from original study
* unable or unwilling to provide written informed consent
* excluded from original study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who underwent an arthroscopic rotator cuff surgery between 2007-2009.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were screened from a large database of 1874 enrolled participants. For the purposes of this project, 90 participants were followed in each arm.
Groups:
- Single-Row Fixation: Single-Row anchor fixation in arthroscopic rotator cuff repair.
- Double-Row Fixation: Double-Row anchor fixation in arthroscopic rotator cuff repair.
Period: Overall Study
Arm/Group | Single-Row Fixation | Double-Row Fixation
Started | 48 | 42
Completed | 43 | 34
Not Completed | 5 | 8
Not completed — Lost to Follow-up | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-Row Fixation | Double-Row Fixation | Total
Number analyzed (Participants) | 43 | 34 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analysis was performed at the 10-year long term follow-up. 5 participants were lost to follow-up in the single row group, and 8 participants were lost to follow-up in the double-row group, and as such were removed from this analysis.
  years | 55.3 (8.2) | 57.2 (6.7) | 56.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analysis was performed at the 10-year long term follow-up. 5 participants were lost to follow-up in the single row group, and 8 participants were lost to follow-up in the double-row group, and as such were removed from this analysis.
  Participants
    Female | 12 | 10 | 22
    Male | 31 | 24 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Analysis was performed at the 10-year long term follow-up. 5 participants were lost to follow-up in the single row group, and 8 participants were lost to follow-up in the double-row group, and as such were removed from this analysis.
  participants
    Canada | 43 | 34 | 77
Affected Shoulder [Number; unit: participants] — Population: Analysis was performed at the 10-year long term follow-up. 5 participants were lost to follow-up in the single row group, and 8 participants were lost to follow-up in the double-row group, and as such were removed from this analysis.
  participants
    Left | 10 | 9 | 19
    Right | 33 | 25 | 58
Tear Size [Mean (Standard Deviation); unit: mm] — Population: Analysis was performed at the 10-year long term follow-up. 5 participants were lost to follow-up in the single row group, and 8 participants were lost to follow-up in the double-row group, and as such were removed from this analysis.
  mm
    Coronal | 21.2 (9.1) | 22.5 (10.7) | 21.8 (9.8)
    Sagittal | 18.8 (7.4) | 18.7 (7) | 18.8 (7.2)
Smoking Status [Count of Participants; unit: Participants] — Population: Analysis was performed at the 10-year long term follow-up. 5 participants were lost to follow-up in the single row group, and 8 participants were lost to follow-up in the double-row group, and as such were removed from this analysis.
  Participants
    Smoker | 7 | 7 | 14
    Nonsmoker | 36 | 27 | 63
Concomitant Biceps Procedure [Count of Participants; unit: Participants] — Population: Analysis was performed at the 10-year long term follow-up. 5 participants were lost to follow-up in the single row group, and 8 participants were lost to follow-up in the double-row group, and as such were removed from this analysis.
  Participants
    No Biceps Procedure | 35 | 25 | 60
    Biceps Tenodesis Procedure | 8 | 9 | 17
Anchors [Median (Inter-Quartile Range); unit: # anchors] — Population: Analysis was performed at the 10-year long term follow-up. 5 participants were lost to follow-up in the single row group, and 8 participants were lost to follow-up in the double-row group, and as such were removed from this analysis.
  # anchors | 1 [1 to 2] | 2 [2 to 3] | 2 [1 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario Rotator Cuff Index
Description: The Western Ontario Rotator Cuff Index (WORC) is a disease specific evaluation, proven to be an accurate and valid assessment of function after. The WORC is a patient-reported measure, 21-question survey. Each question is measured using a visual analog scale rated from 0-100, where higher scores mean better outcome.
Time Frame: 10 year post operative
Measure: Mean (Standard Deviation); unit: score on a scale (0-100)
Arm/Group | Single-Row Fixation | Double-Row Fixation
Number analyzed (Participants) | 43 | 34
score on a scale (0-100) | 72.9 (23.5) | 79.9 (23.4)

2. Secondary Outcome: American Shoulder and Elbow Surgeons Score
Description: The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
Time Frame: 10 year post operative
Measure: Mean (Standard Deviation); unit: units on a scale (0-100)
Arm/Group | Single-Row Fixation | Double-Row Fixation
Number analyzed (Participants) | 43 | 34
units on a scale (0-100) | 80.4 (23.6) | 83.0 (25.1)

3. Secondary Outcome: Constant Score
Description: The Constant Score reflects an overall clinical functional assessment. This instrument is based on a 100-point scoring system. Subjective findings (pain, activities of daily living, and working in different positions) make up a total of 35 points. Objective measurements make up the remaining 65 points.The test is divided into four sub-categories: (1) pain is measured using 4 likert levels (15 points maximum), where a higher score indicates a better outcome; activities of daily living are measured using a likert scale, where a higher number indicates better outcomes (20 points maximum); mobility is measured by an assessor, and rated using a likert scale where a higher score indicates better outcomes (40 points maximum); finally, strength is measured by an assessor where 1 point is given per 0.5kg of force (maximum 25 points), a higher score indicates better outcomes. All categories are added together, and a total score out of 100 is given (higher score indicates better outcome).
Time Frame: 10 year post operative
Population: Not all participants wanted to return to have their strength tested, but agreed to complete questionnaires.
Measure: Mean (Standard Deviation); unit: units on a scale (0-100)
Arm/Group | Single-Row Fixation | Double-Row Fixation
Number analyzed (Participants) | 33 | 28
units on a scale (0-100) | 77.2 (16.7) | 71.3 (25.6)

4. Secondary Outcome: Strength
Description: Strength will be measured using a handheld dynamometer in the abduction position which records kilograms of force. The higher the kilogram of force indicates a better result.
Time Frame: 10 year post operative
Population: Not all participants wanted to return to have their strength tested, but agreed to complete questionnaires.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Single-Row Fixation | Double-Row Fixation
Number analyzed (Participants) | 33 | 28
kg | 7.1 (2.1) | 6.9 (2.7)

ADVERSE EVENTS:
Time Frame: 10 years
Arm/Group | Single-Row Fixation | Double-Row Fixation
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/34
Other Adverse Events (participants affected / at risk) | 0/43 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Row Fixation (N=43) | Double-Row Fixation (N=34)
Revision Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT00253864/Prot_SAP_000.pdf